CLINICAL TRIAL: NCT02031809
Title: Analysis of the Most Common Major Intraoperative Complications During Video-assisted Thoracoscopic Surgery (VATS) Anatomical Resections - On Behalf of MITIG-ESTS
Brief Title: Multicentric Study VATS Major Introperative Complications
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, Datamanager Thoracic Surgery, University Hospital, Gasthuisberg
Other Study IDs: MC_VATS complic
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Lung Neoplasms
Keywords: Thoracic Surgery, Video-Assisted
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No additional unplanned major surgery: uneventfull intra-operative and postoperative course
- Additional unplanned major surgery: Additional per-operative or post-operative unplanned major surgery such as unforeseen pneumonectomy, bilobectomy, lobectomy or additional segmentectomy, repair of major vessels or bronchi, bronchopleural fistula, unplanned surgery to other organs, within 30 days after the primary surgery.
  These do not include:
  * Conversions without additional unplanned major surgery or suddne blood loss less than 500cc
  * Conversions or additional resection for unforeseen oncologic reasons.
  * Plasty, repair or sleeve resection of vessels after deliberate resection or transection for oncologic reasons

SUMMARY:
This study investigates the most common major complications that result in unplanned additional surgery in patients undergoing vats anatomical resections. Several high-volume European centres participate. The purpose is to quantify these major complications, discuss the steps that can be taken to prevent these events, how they can be dealt with, be it by vats or conversion

DETAILED DESCRIPTION:
Vats lobectomy is becoming the standard of care for early stage lung cancer. Several studies have shown feasibility and safety in dedicated centres. Compared to thoracotomy the procedure results in at least equal oncologic results and survival, perhaps better.

Most series do not publish their early experience. They are retrospective and report on lobectomies and segmentectomies, excluding the live-saving pneumonectomies. They are potentially ignoring the intention-to-treat principle, excluding conversions.

Based on scarce existing literature and conference worst-case presentations a pattern of the most common intraoperative major complications can be drawn In Europe, a large percentage of high-volume-centres have now successfully implemented a vats lobectomy program. In this era with low-volume-centres switching into vats anatomical resections, it is important to focus on potentially life-threatening complications. To be aware of potential hazards is the best way to avoid them.

ELIGIBILITY:
Inclusion Criteria:

* Patients that did undergo resection for oncologic reasons

Exclusion Criteria:

* Patients that did not undergo resection for oncologic reasons, such as pleural metastasis, irresectable disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients intended to undergo a vats anatomical resection
Sampling Method: Probability Sample
Enrollment: 3076 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
additional unplanned major surgery | during vats anatomical resection or at revision within 30 days
  the percentage of major complications that resulted in additional unplanned major surgery during vats anatomical resection or at revision within 30 days.

SECONDARY OUTCOMES:
number of conversions to open surgery | during VATS procedure
  The number of VATS procedures that need conversion to open surgery because of major complications or unplanned major surgery

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Dacaluwé, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Dominique Gossot, MD, Principal Investigator — Thoracic Department, Institut Mutualiste Montsouris, 42 Bd Jourdan, F-75014 Paris, France
Locations (9):
- Department of Visceral, Transplant and Thoracic Surgery, Innsbruck University Hospital, Innsbruck, Austria
- Department of Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Denmark
- Thoracic Department, Institut Mutualiste Montsouris, Paris, France
- Katholisches Klinikum, Thoraxchirurgie, Koblenz, Germany
- Division of Thoracic Surgery, Ospedali Riuniti Ancona, Ancona, Italy
- Maatschap Heelkunde Zuid-Limburg, Heerlen, Netherlands
- Karol Marcinkowski University of Med Sciences, Department of Thoracic Surgery, Poznan, Poland
- Department of Thoracic Surgery, A Coruña, Spain
- UniversitätsSpital Zürich, Zurich, Switzerland